CLINICAL TRIAL: NCT02109029
Title: Use of Open-Flow Microperfusion to Measure LY2605541 and Human Insulin Concentrations in Adipose Tissue Interstitial Fluid
Brief Title: A Study of LY2605541 (Insulin Peglispro) and Human Insulin Concentrations in Fat Tissue
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14873; I2R-MC-BIDP (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — basal insulin peglispro; LY2605541; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Peglispro (LY2605541) (Experimental): Part A Cohort 1: (low dose) priming dose (PD) of 2.00 units (U), 0.92 U/hour (U/h) constant infusion of insulin peglispro Part A Cohort 1: (high dose) PD of 8.00 U, 4.50 U/h constant IV infusion of insulin peglispro Part A Cohort 2: (intermediate dose 1) PD of 4.00 U, 1.84/h constant IV infusion of insulin peglispro Part A Cohort 2: (intermediate dose 2) PD of 6.0 U, 2.76 U/h constant IV infusion of insulin peglispro Part B Insulin Peglispro: PD of 6.00 U, 2.76 constant IV infusion of insulin peglispro and a constant infusion of 6 pico moles per kilogram per minute (pmol/kg/min). IV infusion of sinistrin (250 mg/mL, SOC to achieve a steady state for up to 16 hours).
  Interventions: Drug: Insulin Peglispro
- Human Insulin (Active Comparator): Constant IV infusion ( 6 pico moles per kilogram perminute [pmol/kg/min]) of human insulin for up to 36 hours. IV infusion of sinistrin (250 mg/mL, SOC to achieve a steady state for up to 16 hours).
  Interventions: Drug: Human Insulin

INTERVENTIONS:
Drug: Insulin Peglispro — Administered IV
  Other Names: LY2605541
  Arms: Insulin Peglispro (LY2605541)
Drug: Human Insulin — Administered IV
  Arms: Human Insulin

SUMMARY:
LY2605541 is an investigational drug being developed for the treatment of diabetes mellitus. This study is designed to understand how the body handles the investigational drug, and to measure the quantity of LY2605541 in fat tissue. The study has two parts. It involves intravenous (IV) infusion of the investigational drug and a procedure to measure concentrations in the fat tissue. Both parts of the study will be conducted in participants with type 1 diabetes mellitus (T1DM). Part A and B of the study might take up to 7 weeks to complete.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 1 Diabetes Mellitus (T1DM) based on medical history for at least 1 year prior to enrollment
* Have a c-peptide value ≤0.3 nanomoles per liter (nmol/L) at screening
* Have a serum creatinine value within normal limits at screening
* Have a haemoglobin A1c (HbA1c) value ≤75 millimoles per mole (mmol/mol) (9.0%) at screening
* Have a body mass index (BMI) of 20.0-30.0 kilograms per meter squared (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Have known or suspected allergies or hypersensitivities to LY2605541, human insulin, sinistrin, related compounds or any components of the formulations
* Are women who are pregnant or lactating
* Have an abnormal blood pressure for the population as determined by the investigator
* Have renal insufficiency or major renal disorders
* Have proliferative retinopathy or maculopathy
* Have lipodystrophy
* Have any wound healing disorder or are prone to keloid or hypertrophic scar formation
* Have results of screening prothrombin time (PT) and international normalized ratio (INR) tests that are significantly prolonged
* Have a fasting triglycerides value > 4.52 millimoles per liter (mmol/L) (400 milligrams/deciliter (mg/dL))
* Are receiving chronic systemic or inhaled glucocorticoid or have received such therapy within the 4 weeks before dosing
* Have a total daily insulin dose greater than 1.2 units per kilogram (U/kg)
* Regular use or intended use of any over-the-counter or prescription medications or nutritional supplements that affect blood glucose or the body's sensitivity to insulin or that promote weight loss within 14 days prior to dosing
* Regular use or intended use of non-selective beta blockers
* Regular use or intended use of monoamine oxidase (MAO) inhibitors
* Are currently participating in a weight loss program or plan to do so during the course of the study
* Are unwilling to avoid excessive sun exposure, steam baths, saunas, and swimming during the study. Sun cream should be used during sun bathing for the 6-month period following the study
* Are unwilling to avoid extensive consumption of food containing inulin during the study and in the 48-hour period leading up to the clamp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Cohort 1 Insulin Peglispro Low/High: Participants received a priming dose of 2.00 U and 0.92 U/ hour constant intravenous (IV) infusion of insulin peglispro for 36 hours as treatment 1 and received a priming dose of 8.00 U and 4.50/h constant infusion with at least 6 days between doses) as treatment 2.
- Part A: Cohort 1 Insulin Peglispro High/Low: Participants received a priming dose of 8.00 U and 4.50 U/ hour constant intravenous (IV) infusion of insulin peglispro for 36 hours as treatment 1, and an IV priming dose of 2.00 U and 0.92 U/hour constant infusion as treatment 2.
- Part A: Cohort 2 Insulin Peglispro Intermediate Dose 1 and 2: Participants received a priming dose of 4.00 U and 1.84 U/h a constant intravenous (IV) of insulin peglispro for 36 hours as treatment 1, and a 6.00 U priming dose and constant infusion of 2.76U/h of insulin peglispro as treatment 2.
- Part A: Cohort 2 Insulin Peglispro, Intermediate Dose 2 and 1: Participants received a priming dose of 6.00 U and 2.76 U/h constant infusion of insulin peglispro as treatment 1, and 4.00 U and 1.84 U/h constant infusion of insulin peglispro for 36 hours as treatment 2.
- Part B: Insulin Peglispro/Human Insulin: Participant received a priming dose of 6.00 U and 2.76 constant intravenous infusion of insulin peglispro for 36 hours as treatment 1 and 6 pmol/kg/min constant infusion of human insulin as treatment 2.
- Part B: Human Insulin/Insulin Peglispro: Participant received 6 pmol/kg/min constant infusion of human insulin IV as treatment 1 and a priming dose of 6.00 U and 2.76 U/h constant infusion of insulin peglispro and a constant infusion for 36 hours as treatment 2.
Period: Part A
Arm/Group | Part A: Cohort 1 Insulin Peglispro Low/High | Part A: Cohort 1 Insulin Peglispro High/Low | Part A: Cohort 2 Insulin Peglispro Intermediate Dose 1 and 2 | Part A: Cohort 2 Insulin Peglispro, Intermediate Dose 2 and 1 | Part B: Insulin Peglispro/Human Insulin | Part B: Human Insulin/Insulin Peglispro
Started | 2 | 2 | 4 | 4 | 0 | 0
Received One Dose of Study Drug | 2 | 2 | 4 | 4 | 0 | 0
Completed | 2 (Participants from Part A did not move on to Part B.) | 2 (Participants from Part A did not move on to Part B.) | 4 (Participants from Part A did not move on to Part B.) | 4 (Participants from Part A did not move on to Part B.) | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Cohort 1 Insulin Peglispro Low/High | Part A: Cohort 1 Insulin Peglispro High/Low | Part A: Cohort 2 Insulin Peglispro Intermediate Dose 1 and 2 | Part A: Cohort 2 Insulin Peglispro, Intermediate Dose 2 and 1 | Part B: Insulin Peglispro/Human Insulin | Part B: Human Insulin/Insulin Peglispro
Started | 0 | 0 | 0 | 0 | 6 (New participants entered Part B.) | 6 (New participants entered Part B.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Part A Low/High Insulin Peglispro: Participants received 4.00 U priming dose and 1.84 U/h constant IV infusion or 8.00 U priming dose and 4.50 U/h constant IV infusionconstant IV infusion of insulin peglispro for 36 hours with up to 2 weeks between doses.
- Part A Intermediate Insulin Peglispro: Participants received 4.00 U priming dose and 1.84 U/h constant IV infusion or 6.00 U priming dose and 2.76U/h constant IV infusion constant IV infusion of insulin peglispro for 36 hours with up to 2 weeks between doses.
- Part B: Participants first received a priming dose of 8.00 U followed by 2.76 U/h constant intravenous (IV) infusion of LY2605541 for 36 hours or 6 pmol/kg/min constant infusion of human insulin with up to 2 weeks between doses.
- Total: Total of all reporting groups
Arm/Group | Part A Low/High Insulin Peglispro | Part A Intermediate Insulin Peglispro | Part B | Total
Number analyzed (Participants) | 4 | 8 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.2) | 39.0 (7.9) | 40.9 (13.6) | 40.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 3 | 8 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 8 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 8 | 12 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 4 | 8 | 12 | 24
BMI [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m²)] | 27.57 (2.09) | 25.98 (1.87) | 26.73 (1.28) | 26.62 (1.65)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 83.93 (12.63) | 83.80 (8.79) | 83.56 (8.60) | 83.70 (8.93)
HbA1c [Mean (Standard Deviation); unit: percentage of Glycated hemoglobin] | 7.20 (0.88) | 7.51 (0.90) | 7.53 (0.54) | 7.47 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Part B: Pharmacokinetics: Steady-State Concentrations in Adipose Tissue Interstitial Fluid (ISF)
Time Frame: 16, 20, 24, and 28 hours postdose
Population: All participants who received at least 1 dose of study drug in Part B and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol per liter (pmol/L)
Groups:
- Insulin Peglispro: Participants received a priming dose of 2.00 U LY2605541 followed by a constant infusion of 0.92 U/h for up to 36 hours.
- Human Insulin: Participants received 6 pmol/kg/min constant IV infusion of human insulin for up to 36 hours
Arm/Group | Insulin Peglispro | Human Insulin
Number analyzed (Participants) | 10 | 11
picomol per liter (pmol/L) | 11200 (23) | 425 (15)

2. Primary Outcome: Part B: Pharmacokinetics: ISF-to-Serum Concentrations
Description: Absolute concentration of ISF of insulin peglispro and human insulin.
Time Frame: 16, 20, 24, and 28 hours postdose
Population: All participants who received at least 1 dose of study drug in Part B and had evaluable pharmacokinetic data.
Measure: Number; unit: picomol per liter (pmol/L)
Arm/Group | Insulin Peglispro | Human Insulin
Number analyzed (Participants) | 10 | 11
picomol per liter (pmol/L) | 1428.4 | 137.9

ADVERSE EVENTS:
Time Frame: Up to 11 months
Description: All participants received one dose of study drug except one participant did not receive a dose of human insulin.
Groups:
- Part A: Insulin Peglispro 2U: Participants received a priming dose of 2.00 U and 0.92 U/ hour constant intravenous (IV) infusion of insulin peglispro for 36 hours.
- Part A: Insulin Peglispro 4U: Participants received a priming dose of 4.00 U and 4.50 U/ hour constant intravenous (IV) infusion of insulin peglispro for 36 hours.
- Part A: Insulin Peglispro 6U: Participant received a priming dose of 6.00 U and 1.84 constant IV infusion of insulin peglispro respectively, for 36 hours.
- Part A: Insulin Peglispro 8U: Participant received a priming dose of 8.00 U and 2.76 constant IV infusion of insulin peglispro respectively, for 36 hours.
- Part B: Insulin Peglispro: Participant received a priming dose of 6.00 U and 2.76 constant intravenous infusion of insulin peglispro for 36 hours.
- Part B: Human Insulin: Participants received 6 pmol/kg/min constant IV infusion of human insulin for up to 36 hours.
Arm/Group | Part A: Insulin Peglispro 2U | Part A: Insulin Peglispro 4U | Part A: Insulin Peglispro 6U | Part A: Insulin Peglispro 8U | Part B: Insulin Peglispro | Part B: Human Insulin
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/4 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/4 | 3/8 | 1/8 | 0/4 | 4/12 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Insulin Peglispro 2U (N=4) | Part A: Insulin Peglispro 4U (N=8) | Part A: Insulin Peglispro 6U (N=8) | Part A: Insulin Peglispro 8U (N=4) | Part B: Insulin Peglispro (N=12) | Part B: Human Insulin (N=11)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days